CLINICAL TRIAL: NCT01752218
Title: A Single Centre Study to Address Precision and Refractive Predictability of Femtosecond Laser-assisted Astigmatic Keratotomy Following the Cataract Surgery
Brief Title: A Study to Address Precision and Refractive Predictability of Femtosecond Laser-assisted Astigmatic Keratotomy Following the Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technolas Perfect Vision GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1209
Record Dates: First submitted 2012-12-14; First posted 2012-12-19 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Astigmatism
Keywords: Femto-second Laser; arcuate incision; corneal astigmatism; astigmatic keratotomy; Cataract
MeSH Terms: conditions — Astigmatism; Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arcuate Incision (Experimental): Study arm will consist of patients who show cataract and corneal astigmatism.
  Interventions: Device: arcuate incision

INTERVENTIONS:
Device: arcuate incision

SUMMARY:
The purpose of this open, prospective study is to address the effectiveness and precision of the VICTUS™ Femtosecond Laser Platform-assisted astigmatic keratotomy after femtolaser-assisted cataract surgery.

DETAILED DESCRIPTION:
Corneal astigmatism after cataract surgery represents a considerable obstacle in the visual rehabilitation of patients. Up-to-date astigmatic keratotomy represents a standardized and effective procedure that allows decreasing of naturally occurring and surgically induced astigmatism. The shape and architecture of the Arcuate Incisions are pre-calculated based on a particular chosen nomogram. The different parameters of the Arcuate Incisions as radius, opening and position angle and cutting depth can be achieved precisely by the laser technology.

The laser-assisted Cataract surgery and the Arcuate Incisions are performed by means of a femtosecond laser (VICTUS™ FEMTOSECOND LASER PLATFORM®, Technolas Perfect Vision GmbH, Munich, Germany) which is in the presented study under investigation and is already CE-approved.

For this open, prospective data collection several selection criteria have been defined in order to obtain a data set of minimal 43 eyes and maximal 50 eyes. Depending on whether they will be treated unilateral or bilateral the number of subjects enrolled within this study sums up to 22-50 patients. The data is gathered in the Castrop-Rauxel Augenklinik and only from one experienced surgeon.

ELIGIBILITY:
Inclusion Criteria:

* Clear corneal media
* Patients must be at least 40 years of age
* mono- or bilateral Cataract with uncorrected distance visual acuity (UCDVA)

  * 0.63 or glare sensitivity
* Vectorial averaged astigmatism of keratometric and topographic astigmatism:

  * 1.0 D and ≤ 2.0 D
* Patients must have read, understood the Patient Information and signed the informed consent form
* Patients are willing and able to return for follow-up examinations

Exclusion Criteria:

* The maximum K- value may not exceed 60D, the minimal value may not be smaller than 37D
* Pachymetry does not include examination results at an radius of 4.25 mm
* Corneal disease or pathology, such as corneal scaring or opacity, that precludes transmission of laser wavelength or that distorts laser light
* Subjects with a poorly dilating pupil or other defect of the pupil that prevents the iris from adequate retraction peripherally
* Lens/zonular instability such as, but not restricted to, Marfan's Syndrome, Pseudoexfoliation Syndrome, etc.
* Manifest Glaucoma
* Previous intraocular or corneal surgery of any kind, including any type of surgery for either refractive or therapeutic purposes in either eye
* Known sensitivity to planned concomitant medications
* Patients regularly taking medicines that could influence the result of the treatment respectively the vision
* Patients with disorders of the ocular muscle, such as nystagmus or strabismus
* Patients with keratoconus, keratectasia or other irregular cornea changes
* Patients with connective tissue weakness
* Patients who are blind on one eye
* Subjects who are immune compromised or carrying diagnosis of connective tissue disease, clinically significant atopic disease, insulin dependent diabetes mellitus, autoimmune diseases, ocular herpes zoster or simplex, endocrine diseases, lupus, rheumatoid arthritis, collagenosis and other acute or chronic illnesses that will increase the risk to the subject or confound the outcomes of this study.
* Abnormal examination results from slit lamp, fundus examination or IOL Master, age related changes are acceptable
* Patients with eye diseases which decreases the visual acuity such as macular degeneration, macular edema, proliferative diabetic Retinopathy
* Abnormal examination results from Topography, age related changes are acceptable
* Patients who are pregnant or nursing
* Patients with concentration disorders, epilepsy and other complicating diseases
* Patients who are participating in another clinical study 30 days before

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2013-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
subjective cylinder | 3 month postoperative
  At the 3 month visit the subjective cylinder as measured with phoropter or trial frame is ≤ 0.75 D in 60% of the eyes.

SECONDARY OUTCOMES:
topographic corneal cylinder | 3 month postoperative
  At the 3 month visit the value of postoperative corneal astigmatism of the central 3 mm zone, measured with topography, is ≤ 1.0 D in 60% of the eyes
abberrometric corneal astigmatism | 3 month postoperative
  At the 3 month visit the value of postoperative corneal astigmatism of the central 3 mm zone, measured with aberrometry, is ≤ 1.0 D in 60% of the eyes.
keratomic corneal astigmatism | 3 month postoperative
  At the 3 month visit the value of postoperative corneal astigmatism of the central 3 mm zone, measured with keratometry, is ≤ 1.0 D in 60% of the eyes
correction index based on keratometric corneal astigmatism | 3 month postoperative
  At 3 month visit the value of the correction index based on preoperative and postoperative keratometric corneal astigmatism is 0.9+- 0,35 in 70% of the eyes.
correction index based on | 3 month postoperative
  At 3 month visit the value of the correction index based on preoperative keratometric corneal astigmatism and postoperative subjective astigmatism is 0.9+- 0,35 in 70% of the eyes.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hoffmann, Dr., Principal Investigator — Augen- & Laserklinik Castrop-Rauxel GmbH
Locations (1):
- Augen- & Laserklinik Castrop-Rauxel GmbH, Castrop-Rauxel, Germany

REFERENCES:
- [Derived] Wendelstein JA, Hoffmann PC, Schwarzenbacher L, Fischinger IR, Hirnschall N, Menapace R, Langenbucher A, Findl O, Bolz M. Lasting Effects: Seven Year Results of the Castrop Nomogram for Femtosecond Laser-Assisted Paired Corneal Arcuate Incisions. Curr Eye Res. 2022 Feb;47(2):225-232. doi: 10.1080/02713683.2021.1975761. Epub 2021 Sep 7. PMID 34464547
- See also: Sponsor: Technolas Perfect Vision GmbH — http://www.technolaspv.com/
- See also: Investigator's side — http://www.augenklinik-castrop-rauxel.de/